CLINICAL TRIAL: NCT03358797
Title: Community-Based Lifestyle and Leadership Intervention for Primary, Secondary, and Tertiary Prevention of Diabetes in Women in the Arab Community
Brief Title: Community-Based Lifestyle Intervention for Diabetes Prevention in Arab Women
Acronym: CBLI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Donna R Zwas, Director, Linda Joy Pollin Cardiovascular Wellness Center for Women, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 123NDP-HMO-CTIL
Record Dates: First submitted 2017-06-25; First posted 2017-12-02 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Health Behaviors
Keywords: Community-based Intervention; Lifestyle intervention; Diabetes prevention; Leadership; Resilience; Women's health
MeSH Terms: conditions — Diabetes Mellitus; Health Behavior | interventions — Early Growth Response Protein 3

STUDY DESIGN:
Intervention Model Description: Stage 1: interventional, Pre - Post study, with quasi-experimental comparison group Stage 2: interventional, Pre - Post study, with cluster randomization (Pilot study to develop the resiliency training manual will be part of stage 2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- intervention-HPP (Experimental): Community participants will participate in a group-based lifestyle intervention based on the CDC Diabetes Prevention Program, and adapted to the Arabic language, Arab culture, Mediterranean Diet, and adapted to include empowerment, leadership and emotion regulation.
  Interventions: Behavioral: intervention-HPP
- CBLI+RT (Experimental): based on randomization, group that will be assigned to CBLI+RT will receive the CBLI curriculum (as described in the intervention-HPP arm) in addition to the resiliency training
  Interventions: Behavioral: Community based intervention with resilience training
- Attention control (CBLI-) (Experimental): The attention control group will receive the core curriculum of the CBLI (as described in the intervention-HPP arm) only without the resiliency training. The sessions of the resiliency training will be replaced with sessions on health topics that do not contribute to our outcome (increased resiliency) (i.e. breast cancer, osteoporosis)
  Interventions: Behavioral: Attention-control
- Pilot (Experimental): This group will not be randomized. The group will receive the CBLI content (as described in the intervention-HPP arm) in addition to the resiliency training. The aim of this pilot is to create a resiliency training manual to be implemented in the following groups that will be assigned to receive the CBLI+RT
  Interventions: Behavioral: Pilot

INTERVENTIONS:
Behavioral: Attention-control — Lifestyle intervention with presentations by multiple professionals (nutritionists, exercise trainers, and psychotherapists), this intervention will include Mediterranean diet education, physical activity, social support, food tasting and cooking, goal setting,and women's health topics
  Arms: Attention control (CBLI-)
Behavioral: Community based intervention with resilience training — Lifestyle intervention with presentations by multiple professionals (nutritionists, exercise trainers, and psychotherapists), this intervention will include Mediterranean diet education, physical activity, social support, food tasting and cooking, goal setting, and women's health topics. In addition, there will be content targeting resilience training including: positive emotions, cognitive flexibility, life meaning, and active coping strategies.
  Arms: CBLI+RT
Behavioral: intervention-HPP — Lifestyle intervention with presentations by multiple professionals (nutritionists, exercise trainers, and psychotherapists), this intervention will include Mediterranean diet education, physical activity, social support, food tasting and cooking, goal setting,and women's health topics. In addition, there will be training in leadership skills, community interventions, community needs assessment, intervention planning and outcomes assessment.
  Arms: intervention-HPP
Behavioral: Pilot — Lifestyle intervention with presentations by multiple professionals (nutritionists, exercise trainers, and psychotherapists), this intervention will include Mediterranean diet education, physical activity, social support, food tasting and cooking, goal setting, and women's health topics. In addition, there will be content targeting resilience training including: positive emotions, cognitive flexibility, life meaning, and active coping strategies.
  Arms: Pilot

SUMMARY:
Arab women present increased risk for diabetes, with a 70% greater risk for adult-onset diabetes and a significantly younger age at onset compared with Jewish Israelis. In fact, the rate of diabetes for Arab women in Jerusalem is 4 times higher compared with their Jewish counterparts. Group lifestyle interventions such as the Diabetes Prevention Program (DPP) have documented effectiveness in preventing diabetes; however, many fail to demonstrate outcome maintenance. We predict that integrating leadership skills training into the gold standard DPP would improve the long-term outcome maintenance.

Stage 1: A pre-post study design will be utilized, where all community participants will be exposed to intervention components. The sample was selected from pre-existing groups in the local community center, based on their leadership potential.

phase 2: The second stage of the trial will not include the leadership component, but instead it will incorporate resiliency training and it aims to evaluate the effect of increased resiliency on the main outcomes including improvement in healthy behaviors such as adherence to Mediterranean diet and as well as a reduction in sedentary lifestyle and increased engagement in physical activity. In addition, resiliency training is likely to improve the maintenance of these behaviors.

DETAILED DESCRIPTION:
The purpose of this study is to design, implement and evaluate a community based lifestyle intervention that integrates a leadership skills training for Palestinian women living in East Jerusalem.

Stage 1: A pre-post study design will be utilized, where all community participants will be exposed to intervention components. The sample was selected from pre-existing groups in the local community center, based on their leadership potential. The Community-Based Lifestyle Intervention (CBLI) was developed by integrating leadership skill training to the gold standard Diabetes Prevention Program (DPP). According to social cognitive theory, engaging in lay leadership can help maintain health behaviors by providing leaders with social support, behavioral reinforcement, outcome expectancies, reciprocal determinism, and building self-efficacy. Fostering social change and empowering individuals, mobilizing community members is also an effective, low cost method for widespread impact on health behavior and health outcomes within the members' community. This is particularly true for women and minority populations. All intervention components were adapted to the specific culture, language, gender, and religious sensitivities of Palestinian female society.

The program will consist of 22 sessions presented by multiple professionals (nutritionists, exercise trainers, health coaches, and psychotherapists). Session content includes Mediterranean diet education, social support, food tasting and cooking, goal setting, self-monitoring, planning, conscious eating, leadership and lay leader training, initiative-taking, group dynamics, project design, community needs assessment, and project evaluation. The study is implemented in partnership with local community centers.

It is hypothesized that Arab women who participate in this community intervention will have improved - and maintained- healthy eating behaviors (i.e. Mediterranean Diet), reduced unhealthy eating behaviors (i.e. Western diet), increased engagement in physical activity and reduced risk of obesity (weight, BMI).

The second stage of the trial will not include the leadership component, but instead it will incorporate resiliency training and it aims to evaluate the effect of increased resiliency on the main outcomes including improvement in healthy behaviors such as adherence to Mediterranean diet and as well as a reduction in sedentary lifestyle and increased engagement in physical activity. In addition, resiliency training is likely to improve the maintenance of these behaviors.

Resiliency can be defined as a personal trait that contributes to the individual's ability to recover from stressful events. It is the ability to achieve, retain, or regain a level of physical or emotional health after illness or loss (bounce back). This characteristic is also considered a protective strength against mental problems, and the ability to effectively adapt to changes and recover from stressful events. Psychological stress is associated with increased risk of non-communicable diseases pose the greatest burden to public health, including heart disease. Additionally, people experiencing psychosocial challenges like isolation and life stress, are found to be less physically active, which is considered an independent risk factor for heart disease. Therefore, effective interventions that aim to reduce stress and anxiety and improve social connectedness are potential means of preventing and managing chronic diseases.

The present study (stage 2) will employ a cluster-randomized trial in which community centers will be assigned to either intervention group or attention control group. The intervention group will receive the CBLI content curriculum (as described above) in addition to the resiliency training (hence CBLI+RT). The attention control group will receive the core curriculum of the CBLI (CBLI-) only without the resiliency training. The sessions of the resiliency training will be replaced with sessions on health topics that do not contribute to our outcome (increased resiliency).

All intervention components were adapted to the specific culture, language, gender, and religious sensitivities of Palestinian female society.

It is hypothesized that Arab women who participate in this community intervention will have improved - and maintained- healthy eating behaviors (i.e. Mediterranean Diet), reduced unhealthy eating behaviors (i.e. Western diet), increased engagement in physical activity and reduced risk of obesity (weight, BMI).

The integration of positive psychology which focuses on individual's strengths through the resiliency training in the second stage of this trial, is hypothesized to be associated with improving-and maintain- healthy behaviors such as healthy diet, increased engagement in physical activity, and reducing unhealthy behaviors such as the consumption of western diet.

The first group will be assigned as a pilot study. This group will not be randomized but will receive the CBLI+RT in order to develop a resiliency training manual to be implemented in the following groups that will be assigned to receive RT in addition to the CBLI core curriculum.

ELIGIBILITY:
Inclusion Criteria:

* Over age 18
* Able to commit to the intervention timetable

Exclusion Criteria:

* Younger than age 18
* Unable to commit to the intervention timetable
* Were not pregnant with expected delivery during the intervention
* Were suffering from other serious mental or physical illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-12-29 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Mediterranean Diet adherence | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be assessed through Panagiotakos' Mediterranean Diet score (an 11 item self-report measure of adherence to the Mediterranean food pattern) which was adapted to Israeli diet and the Arab culture. Items assessing potato and alcohol consumption were removed and an item assessing nut consumption was added
Change in physical activity engagement | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be assessed through self report of minutes engaged in vigorous and moderate physical via questionnaires.

SECONDARY OUTCOMES:
Change in Plasma levels of Hemoglobin A1c (HbA1c) | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of Hemoglobin A1c (HbA1c)
Change in Plasma levels of total cholesterol | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of total cholesterol
Change in Plasma levels of HDL | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of HDL
Change in Plasma levels of LDL | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of LDL
Change in Plasma levels of triglycerides | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  The participants will be referred to their national health insurance in order to conduct a blood test for plasma levels of triglycerides
Change in Body Mass Index (BMI) | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  BMI will be calculated by measuring weight and height for each participant.
Change in Blood Pressure (BP) | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be measured using standard procedures with an electronic BP apparatus and the recorded measurement is the average of 2 measurements taken in the seated position
Change in Cardiovascular Disease Knowledge | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be assessed through self report questionnaire based on the American Heart Association's knowledge survey items
Stages of Change for targeted health behaviors | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be assessed through self report questionnaire
Change in Leadership Self-Efficacy | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Will be assessed through self report questionnaire
Change in Resilience | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Resilience will be measured through the validated 10 items Connor-Davidson Resilience Scale (CD-RISC-10)
Change in Sense of Coherence | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Sense of coherence will be measured through the Sense of Coherence 13-item scale
Change in Self-Rated health | Baseline, 6 months after intervention initiation and 6 months following project completion (1 year later)
  Self reported status of health will be measured using the Self-Rated health questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Donna Zwas, MD, MPH, Principal Investigator — Hadassah University Medical Center
Locations (1):
- Beit-Safafa community center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Undecided
yes, to investigators with certified GCP upon request

REFERENCES:
- [Background] Anderson ES, Winett RA, Wojcik JR. Self-regulation, self-efficacy, outcome expectations, and social support: social cognitive theory and nutrition behavior. Ann Behav Med. 2007 Nov-Dec;34(3):304-12. doi: 10.1007/BF02874555. PMID 18020940
- [Background] Lorig KR, Mazonson PD, Holman HR. Evidence suggesting that health education for self-management in patients with chronic arthritis has sustained health benefits while reducing health care costs. Arthritis Rheum. 1993 Apr;36(4):439-46. doi: 10.1002/art.1780360403. PMID 8457219
- [Background] Heath GW. The role of the public health sector in promoting physical activity: national, state, and local applications. J Phys Act Health. 2009 Nov;6 Suppl 2:S159-67. PMID 20120125
- [Background] Kim K, Choi JS, Choi E, Nieman CL, Joo JH, Lin FR, Gitlin LN, Han HR. Effects of Community-Based Health Worker Interventions to Improve Chronic Disease Management and Care Among Vulnerable Populations: A Systematic Review. Am J Public Health. 2016 Apr;106(4):e3-e28. doi: 10.2105/AJPH.2015.302987. Epub 2016 Feb 18. PMID 26890177
- [Background] Koniak-Griffin D, Brecht ML, Takayanagi S, Villegas J, Melendrez M, Balcazar H. A community health worker-led lifestyle behavior intervention for Latina (Hispanic) women: feasibility and outcomes of a randomized controlled trial. Int J Nurs Stud. 2015 Jan;52(1):75-87. doi: 10.1016/j.ijnurstu.2014.09.005. Epub 2014 Sep 22. PMID 25307195
- [Background] Walton JW, Snead CA, Collinsworth AW, Schmidt KL. Reducing diabetes disparities through the implementation of a community health worker-led diabetes self-management education program. Fam Community Health. 2012 Apr-Jun;35(2):161-71. doi: 10.1097/FCH.0b013e31824651d3. PMID 22367263
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Panagiotakos DB, Pitsavos C, Stefanadis C. Dietary patterns: a Mediterranean diet score and its relation to clinical and biological markers of cardiovascular disease risk. Nutr Metab Cardiovasc Dis. 2006 Dec;16(8):559-68. doi: 10.1016/j.numecd.2005.08.006. Epub 2006 Feb 9. PMID 17126772
- [Background] The National Diabetes Registry (Total Population). (n.d.). Retrieved from https://www.health.gov.il/English/MinistryUnits/ICDC/disease_Registries/Pages/diabetes_reg.aspx.
- [Background] Diabetes Prevention Program (DPP) Research Group. The Diabetes Prevention Program (DPP): description of lifestyle intervention. Diabetes Care. 2002 Dec;25(12):2165-71. doi: 10.2337/diacare.25.12.2165. PMID 12453955
- [Background] Idler EL, Angel RJ. Self-rated health and mortality in the NHANES-I Epidemiologic Follow-up Study. Am J Public Health. 1990 Apr;80(4):446-52. doi: 10.2105/ajph.80.4.446. PMID 2316767
- [Background] Eriksson M, Mittelmark MB. The Sense of Coherence and Its Measurement. 2016 Sep 3. In: Mittelmark MB, Sagy S, Eriksson M, Bauer GF, Pelikan JM, Lindstrom B, Espnes GA, editors. The Handbook of Salutogenesis [Internet]. Cham (CH): Springer; 2017. Chapter 12. Available from http://www.ncbi.nlm.nih.gov/books/NBK435830/ PMID 28590637
- [Background] Cheng C, Dong D, He J, Zhong X, Yao S. Psychometric properties of the 10-item Connor-Davidson Resilience Scale (CD-RISC-10) in Chinese undergraduates and depressive patients. J Affect Disord. 2020 Jan 15;261:211-220. doi: 10.1016/j.jad.2019.10.018. Epub 2019 Oct 12. PMID 31654919